CLINICAL TRIAL: NCT05525416
Title: Sex Differences in Sympathetic Vascular Reactivity at High Altitude
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00096808
Record Dates: First submitted 2022-07-22; First posted 2022-09-01 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-03

CONDITIONS: Vasodilation; Vasoconstriction
MeSH Terms: conditions — Aneurysm | interventions — Nitroprusside; Phenylephrine; Norepinephrine; Propranolol; Phentolamine

STUDY DESIGN:
Intervention Model Description: Participants will partake in both arms of the study, which include: 1) low altitude and 2) high altitude assessments.
Masking Description: Due to the study design, masking is not possible. The time points and dosages of the study drug will be known to the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Altitude (Experimental): Participants will be assessed at an altitude of <1050m.
  Interventions: Drug: Sodium Nitroprusside; Drug: Phenylephrine Hydrochloride; Drug: Norepinephrine; Other: Isometric Handgrip and Post-Exercise Circulatory Occlusion; Other: Rhythmic Handgrip; Other: Cold Pressor Test; Drug: Propranolol Hydrochloride; Drug: Phentolamine Mesylate
- High Altitude (Experimental): Participants will be assessed on a high-altitude expedition at an elevation of 3,800m.
  Interventions: Drug: Sodium Nitroprusside; Drug: Phenylephrine Hydrochloride; Drug: Norepinephrine; Other: Isometric Handgrip and Post-Exercise Circulatory Occlusion; Other: Rhythmic Handgrip; Other: Cold Pressor Test; Drug: Propranolol Hydrochloride; Drug: Phentolamine Mesylate

INTERVENTIONS:
Drug: Sodium Nitroprusside — A bolus injection of sodium nitroprusside will be given to lower blood pressure and evaluate baroreflex function.
Drug: Phenylephrine Hydrochloride — A bolus injection of phenylephrine will be given to raise blood pressure and evaluate baroreflex function immediately following the sodium nitroprusside infusion.
  Other Names: Neo-Synephrine
Drug: Phenylephrine Hydrochloride — Investigators will give three incremental doses via brachial artery catheter to observe α1-adrenoreceptor mediated vasoconstriction. This will occur three times throughout the protocol.
Drug: Norepinephrine — Investigators will give three incremental doses via brachial artery catheter to observe adrenoreceptor activation. This will occur three times throughout the protocol.
Other: Isometric Handgrip and Post-Exercise Circulatory Occlusion — Participants will perform 2 minutes of isometric handgrip at 30% maximal voluntary contraction followed by 2 minutes of post-exercise circulatory occlusion to assess the reactivity of the blood vessels to exercise and the metaboreflex.
Other: Rhythmic Handgrip — Participants will perform 3 minutes of rhythmic handgrip at 25% maximal voluntary contraction to assess the reactivity of blood vessels to dynamic exercise.
Other: Cold Pressor Test — Standardized sympathetic stressor involving submersion of the hand in ice-cold water for 3-minutes, aiming to elicit endogenous neurotransmitter release and blood pressure increases.
Drug: Propranolol Hydrochloride — Local infusion via brachial artery catheterization will occur continuously for the remainder of the study. Propranolol is a beta-adrenergic antagonist and will allow investigation of the role of beta receptors in responses to various stressors. The above phenylephrine, norepinephrine, isometric handgrip, post-exercise circulatory occlusion, and rhythmic handgrip protocols will be repeated under propranolol infusion.
Drug: Phentolamine Mesylate — Local infusion via brachial artery catheterization will occur continuously for the remainder of the study. Phentolamine is an alpha-adrenergic antagonist and will allow investigation the role of alpha receptors in responses to various stressors. It will be continuously infused with propranolol. The above phenylephrine, norepinephrine, isometric handgrip, post-exercise circulatory occlusion, and rhythmic handgrip protocols will be repeated under propranolol infusion.

SUMMARY:
This study aims to investigate sex differences in blood pressure control associated with exposure to acute hypoxia (low oxygen), and short term acclimatization to hypoxia at high altitude.

DETAILED DESCRIPTION:
About 200 million people worldwide live at high altitudes and millions of others travel to high altitude every year for work or pleasure. At high altitude participants are exposed to a lower than normal level of oxygen, also known as hypoxia. This causes stress to the human body, which will adapt in order to maintain adequate oxygen delivery to its tissues. One of these adaptations is an increase in activity of participants' sympathetic nervous system ("fight or flight" response). Sympathetic nerve activity affects the size of participants' blood vessels, which in turn will affect blood pressure. Men and women regulate their blood pressure in different ways; for example, women tend to have lower blood pressure and sympathetic nerve activity than men. Women also appear to have less constriction of their blood vessels in response to stress. This may be in part because estrogen causes blood vessels to dilate. It may also be due to differences in the receptors which are activated by the sympathetic nervous system. These receptors are called alpha and beta receptors and respond to sympathetic nerve activity in opposite directions. Women represent 50% of the population living at and travelling to high altitude, therefore, it is important to understand the differences in how men and women respond to low oxygen.

The main purpose of this study is to examine the differences between men and women in the sympathetic nervous system control of blood vessels during exposure to low oxygen. To study this question, the investigators will test how blood vessels respond to stressors in both men and women. Participants will be recruited at the Canadian sites, and the investigators will test them while they breathe low oxygen for a short amount of time at low altitude. The investigators will also perform assessments on the same participants during a two week stay at high altitude at White Mountain, CA, which is at an altitude of 3,800m. These data will have implications in the basic understanding of differences between male and female physiology. Specifically, to males and females living or travelling to high altitude.

ELIGIBILITY:
Inclusion Criteria:

* Between ages of 18-50
* No medical history of cardiovascular, respiratory, nervous system, or metabolic disease
* Females must be pre-menopausal

Exclusion Criteria:

* Any known cardiovascular, respiratory, nervous system, or metabolic disease (however, participants with controlled arterial hypertension will not be excluded)
* Having travelled above 2,000m within 1 month of testing at low and high altitude
* Females who are pregnant, confirmed by a pregnancy test
* Females who are post-menopausal
* Participants that are classified as obese (body mass index > 30kg⋅m²)
* Participants who are current daily smokers
* Those with a known allergy to sulfites
* Participants taking monoamine oxidase (MAO) inhibitors or tricyclic antidepressants or other medications that have contraindications with the study drugs
* Participants who are still within the washout period from participating in other studies involving drugs.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2022-07-28 (Actual); Primary Completion 2023-02-05 (Actual); Study Completion 2023-02-05 (Actual)

PRIMARY OUTCOMES:
Change in systolic, diastolic, and mean arterial blood pressure | 3 minutes
  modified oxford
Change in arterial blood flow | 1 hour 30 minutes
  phenylephrine and norepinephrine sensitivity
Change in vascular conductance | 20 minutes
  exercise and metaboreflex reactivity
Cold pressor test | 3 minutes
  sympathetic reactivity
Propranolol | 2 hours
  changes in vascular conductance
Phentolamine | 1 hour
  changes in vascular conductance

CONTACTS AND LOCATIONS:
Overall Officials: Sean van Diepen, MD, MSc, Principal Investigator — University of Alberta; Craig D Steinback, PhD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia - Okanagan, Kelowna, British Columbia

REFERENCES:
- [Background] Hart EC, Charkoudian N, Wallin BG, Curry TB, Eisenach JH, Joyner MJ. Sex differences in sympathetic neural-hemodynamic balance: implications for human blood pressure regulation. Hypertension. 2009 Mar;53(3):571-6. doi: 10.1161/HYPERTENSIONAHA.108.126391. Epub 2009 Jan 26. PMID 19171792
- [Background] Mazzeo RS, Child A, Butterfield GE, Mawson JT, Zamudio S, Moore LG. Catecholamine response during 12 days of high-altitude exposure (4, 300 m) in women. J Appl Physiol (1985). 1998 Apr;84(4):1151-7. doi: 10.1152/jappl.1998.84.4.1151. PMID 9516178
- [Background] Purdy GM, James MA, Rees JL, Ondrus P, Keess JL, Day TA, Steinback CD. Spleen reactivity during incremental ascent to altitude. J Appl Physiol (1985). 2019 Jan 1;126(1):152-159. doi: 10.1152/japplphysiol.00753.2018. Epub 2018 Nov 21. PMID 30462566
- [Background] Usselman CW, Gimon TI, Nielson CA, Luchyshyn TA, Coverdale NS, Van Uum SH, Shoemaker JK. Menstrual cycle and sex effects on sympathetic responses to acute chemoreflex stress. Am J Physiol Heart Circ Physiol. 2015 Mar 15;308(6):H664-71. doi: 10.1152/ajpheart.00345.2014. Epub 2014 Dec 19. PMID 25527774